CLINICAL TRIAL: NCT00607542
Title: Pediatric Pharmacokinetic and Pharmacodynamic Study of Oral Baclofen for the Treatment of Spasticity Associated With Cerebral Palsy
Brief Title: Oral Baclofen Pharmacokinetics and Pharmacodynamics in Children With Spasticity
Acronym: Best PK/PD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NICHD-2005-13-2; 267200603421
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-02

CONDITIONS: Spasticity; Cerebral Palsy
Keywords: spasticity; cerebral palsy; baclofen; pharmacokinetics; pharmacodynamics; dosing; safety; efficacy
MeSH Terms: conditions — Muscle Spasticity; Cerebral Palsy | interventions — Baclofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Active Comparator): starting dose of baclofen 2.5 mg PO TID with dose escalation as tolerated
  Interventions: Drug: baclofen

INTERVENTIONS:
Drug: baclofen — 2.5 mg oral baclofen tablets given three times a day; dose gradually escalated as specified in the protocol
  Other Names: Lioresal

SUMMARY:
Oral baclofen is used commonly to treat spasticity in children with cerebral palsy. Although for adults there is dosing,safety and efficacy information in the package insert, this is not the case for children. The purpose of this study is to determine how fast the drug is cleared from the body, the correct dose, and long-term safety and efficacy for children with spasticity.

DETAILED DESCRIPTION:
Although oral baclofen has been used for several decades for the treatment of spasticity in adults and in children, there is very little data regarding the pharmacokinetic (PK) or pharmacodynamic (PD) properties of baclofen in children. Therefore, pediatric guidelines, including dose ranges, dosing schedules, dose escalation strategies and anticipated side effects are extrapolated from adult data and require an assumption that safety and efficacy in children is comparable to that in adults. Furthermore, there is wide variability in dosing strategies among practitioners who treat children with cerebral palsy (CP) with respect to starting doses, maximum doses and rates of dose escalation.Establishment of safe and effective dosing strategies for children with CP requires an understanding of the PK and PD properties of baclofen in children and recognition of individual differences that may contribute to divergent clinical responses to baclofen among children with CP.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 2-16 years, inclusive.
2. Triceps skinfold thickness between the 5th and 95th percentiles for age (Refer to Appendix 3).
3. Gross Motor Function Classification Scale (GMFCS) Level II - V (GMFCS classifies children by functional mobility with Level I indicating minimal motor disability and V indicating total body involvement and dependence on others for mobility (Palisano et al, 1997).
4. Ashworth score of 2 or higher in at least one arm and one leg (knee + elbow flexors and/or extensors).
5. Cerebral Palsy: Motor disability due to a static, non-progressive brain injury/ malformation occurring prenatally or any time prior to the age of 2 years.
6. No history of baclofen use within the past 4 months.
7. Female subject, is premenarchal, or is incapable of pregnancy because of a hysterectomy or tubal ligation; or female subject who is sexually active and capable of pregnancy, has been using an acceptable method of contraception (hormonal contraceptives, intrauterine device, spermicide and barrier) for at least one month prior to study entry and agrees to continue to use one of these for the duration of the study; or female subject who is sexually abstinent and capable of pregnancy, agrees to continued abstinence or to use an acceptable method of birth control (either intrauterine device or spermicide and barrier) should sexual activity commence.
8. Subject ≥10 years of age has negative urine tests at screening and baseline for alcohol, non-medically prescribed drugs of abuse, and no history of tobacco use.

Exclusion Criteria:

1. Hypersensitivity to baclofen.
2. Selective dorsal rhizotomy.
3. Active intrathecal baclofen pump within the past 6 months.
4. Use of botulinum toxin in past 4 months or use any time during the study.
5. Use of tone altering medications (e.g. baclofen, benzodiazepines, levodopa, trihexyphenidyl) for >3 consecutive days duration within the past 4 months.
6. Start of any drug or product known to be a significant cytochrome P450 enzyme inducer or inhibitor within the past 30 days.
7. Orthopaedic surgery within the past year or any time during the study.
8. Abdominal surgery within the past six months or any time during the study.
9. Uncontrolled seizures (baseline seizure frequency >1 per month or history of more than 2 prolonged seizures lasting longer than 5 minutes duration within the past year.
10. Severe behavior difficulties or psychiatric disturbance
11. Proven gastric dysmotility: known history of abnormal gastric emptying study and/or history of vomiting 3 or more times per week.
12. Severe Gastroesophageal Reflux Disease: known history of esophagitis (documented on abnormal endoscopy or biopsy).
13. Malnutrition: defined as triceps skin fold thickness less than 5th or greater than 95th percentile for age.
14. Renal or Liver disease: Elevated bilirubin, LFTs greater than twice the upper limit of normal, reduced BUN/Cr ratio (<5), or abnormal creatinine clearance that is clinically significant as determined by the investigator.
15. Abnormal CBC: Anemia, polycythemia, neutropenia, leukocytosis, thrombocytopenia, or thrombocytosis clinically significant as determined by the investigator.
16. Pregnancy or lactation.
17. Severe respiratory or cardiac disease: Requirement for prolonged supplemental oxygen (>7 days), history of clinically significant congenital heart disease, congestive heart failure or cardiomegaly, and/or hospital admission within past 6 months for cardiac symptoms or respiratory distress.
18. Previous baclofen failure: Lack of response to baclofen or presence of unacceptable side effects. If previous baclofen therapy was tried >4 months prior to study and discontinued, the decision to enroll subject will be at the discretion of the site investigator and reason for discontinuation of oral baclofen will be recorded.
19. Use of medications that interfere with measurements of serum creatinine levels within the past 14 days (e.g., trimethoprim-sulfa, fibric acid derivatives other than gemfibrizol, keto acids, salicylates, some cephalosporins, cimetidine, phenacemide) .
20. Subject tests positive at screening for the hepatitis B surface antigen or hepatitis C antibody, or has a history of a positive result for one of these tests.
21. Subject is known to have tested seropositive for the human immunodeficiency virus (HIV) or subject is concomitantly receiving anti-retroviral therapy.
22. Any serious, unstable medical illness or clinically significant abnormal laboratory assessment that would adversely impact the scientific interpretability or unduly increase the risks of the protocol.
23. Subject has a disorder or history of a condition, other than that related to CP that could interfere with drug absorption, distribution, metabolism, or excretion.
24. Any condition which would make the patient

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2008-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Determine pharmacokinetic parameters of oral baclofen in children with spasticity associated with cerebral palsy (CP). | 1 year
Describe the relationship between plasma concentrations of oral baclofen and clinical measures of spasticity. | 1 year
Determine optimal dosing range and interval for administration of oral baclofen for use in a randomized clinical trial of safety and efficacy. | 1 year

SECONDARY OUTCOMES:
Describe the relationship between plasma concentrations of oral baclofen and measures of strength, function, ease of care, pain/comfort and health related quality of life. | 1 year
Describe the safety and tolerability of oral baclofen in children with spasticity associated with CP. | 1 year
Investigate preliminarily whether oral baclofen improves dystonia | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Janice Brunstrom, MD, Principal Investigator — Washington University of St. Louis; Richard Stevenson, MD, Principal Investigator — University of Virginia
Locations (11):
- United States (11):
  - Rehabilitation Institute of Chicago, Chicago, Illinois
  - Children's Hospital of Lousiana, New Orleans, Louisiana
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Gillette Children's Speciality Healthcare, Saint Paul, Minnesota
  - Children's Mercy Hospital and Clinics, Kansas City, Missouri
  - Washington Univeristy - St. Louis Children's hospital, St Louis, Missouri
  - SUNY Upstate Medical University, Syracuse, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Texas Children's Hospital, Houston, Texas
  - Kluge Children's Rehabilitation Center - University of Virginia, Charlottesville, Virginia
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Derived] McLaughlin MJ, He Y, Brunstrom-Hernandez J, Thio LL, Carleton BC, Ross CJD, Gaedigk A, Lewandowski A, Dai H, Jusko WJ, Leeder JS. Pharmacogenomic Variability of Oral Baclofen Clearance and Clinical Response in Children With Cerebral Palsy. PM R. 2018 Mar;10(3):235-243. doi: 10.1016/j.pmrj.2017.08.441. Epub 2017 Sep 1. PMID 28867665
- [Derived] He Y, Brunstrom-Hernandez JE, Thio LL, Lackey S, Gaebler-Spira D, Kuroda MM, Stashinko E, Hoon AH Jr, Vargus-Adams J, Stevenson RD, Lowenhaupt S, McLaughlin JF, Christensen A, Dosa NP, Butler M, Schwabe A, Lopez C, Roge D, Kennedy D, Tilton A, Krach LE, Lewandowski A, Dai H, Gaedigk A, Leeder JS, Jusko WJ. Population pharmacokinetics of oral baclofen in pediatric patients with cerebral palsy. J Pediatr. 2014 May;164(5):1181-1188.e8. doi: 10.1016/j.jpeds.2014.01.029. Epub 2014 Mar 5. PMID 24607242